CLINICAL TRIAL: NCT05237024
Title: Monitoring of Physiologic Changes Associated With Immune System Activation Associated With Vaccination Against the SARS-CoV-2 Virus: Vaccine-Induced Inflammation Identification
Brief Title: (VIII): The Eight Study and Immunologic Response Sub-study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: physIQ, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CTP-024
Record Dates: First submitted 2021-12-29; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Vaccine Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physiology Monitoring: The study's objective is to test the hypothesis that immune system activation and subsequent systemic inflammation can be detected through continuously tracking multiple bio signals including physiologic variables (ECG, skin temperature and their derivatives) and behavioral variables (activity and sleep from accelerometers) collected during routine activities of daily living using wearable biosensors.
- Physiology & Immune Monitoring: A limited sub-study including 30 individuals enrolled in the primary study (not retrospective group) will incorporate serial blood draws relative to the vaccine doses. The purpose of the serologies and immunoassays is to explore the correlation an individual's development of a vaccine-induced immune response with changes in the continuous physiologic data surrounding the immunization process.

SUMMARY:
The study's objective is to test the hypothesis that immune system activation and subsequent systemic inflammation can be detected through continuously tracking multiple bio signals including physiologic variables (ECG, skin temperature and their derivatives) and behavioral variables (activity and sleep from accelerometers) collected during routine activities of daily living using wearable biosensors. In the sub-study, the objective is to explore the association between these objectively measured physiologic changes and vaccine-induced humoral and T-cell responses.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 years of age or older.
* Is able to speak and read English.
* Plan to receive either the Moderna or Pfizer vaccine (mRNA vaccine).
* No known prior COVID-19 infection.

Exclusion Criteria:

* Known allergy to the adhesive used on the VitalPatch.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults that plan to receive COVID-19 vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Collect bio signal data before and after vaccination in ~100 individuals using one or more wearable biosensors. | December, 2022
Evaluate the relationship between the MCI and individual bio signals parameters and the subjective symptoms experienced by participants. | December, 2022
Explore the association between these objectively measured physiologic changes and vaccine-induced humoral and T-cell responses. | December, 2022

CONTACTS AND LOCATIONS:
Overall Officials: Steve Steinhubl, MD, Principal Investigator — CMO
Locations (2):
- physIQ, Chicago, Illinois, United States
- Cell Carta, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No